CLINICAL TRIAL: NCT01300884
Title: Sierra High Definition Ano-Rectal Manometry
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Other Study IDs: 200705716
Record Dates: First submitted 2011-01-19; First posted 2011-02-23 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Constipation; Fecal Incontinence
MeSH Terms: conditions — Constipation; Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- healthy volunteers
- patients with fecal incontinence
- patients with constipation

SUMMARY:
Hypotheses: High definition manometry (HDM) is safe and feasible in humans; HDM accurately characterizes anorectal anatomy and function in healthy humans; HDM provides comparable information regarding the structure and function of the anorectal region, to that obtained from ano-rectal manometry and anal ultrasonography (AUS), in patients with fecal incontinence or constipation.

Methods: 20 healthy volunteers, 20 patients with fecal incontinence, 20 patients with constipation will be recruited. Because anorectal disorders are more common in women, the investigators will recruit approximately 8 men and 12 women in each group. Each subject will undergo anorectal manometry, anal ultrasound and high definition manometry.

Data Analysis: Spearman correlational analysis will be performed to compare the parameters listed above. Also, the diagnostic yield of anal ultrasonography vs HDM in identifying anatomic sphincter defects will be assessed.

ELIGIBILITY:
Inclusion Criteria:

For patients:

1. Either fecal incontinence (the occurrence of at least one episode of involuntary discharge of stool matter per week) or constipation (Rome III criteria) (16,17)
2. Adults between the ages of 18-80 yrs.

For healthy volunteers:

1. Adults between the ages of 18-80 yrs
2. No gastrointestinal symptoms

Exclusion Criteria:

1. Rectal prolapse or anal fissure on physical examination
2. Recent pelvic or recto-anal surgery (< 6 months ago)
3. History of pelvic irradiation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit 20 healthy volunteers, 20 patients with fecal incontinence, 20 patients with constipation. Because anorectal disorders are more common in women, we will recruit approximately 8 men and 12 women in each group. Because it is possible subjects may sign consent but not participate in the study, or drop out of the study before completion, we will recruit a total of 80 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of HDM in three groups of human subjects; healthy humans, patients with fecal incontinence and patients with chronic constipation | One visit

CONTACTS AND LOCATIONS:
Overall Officials: Satish SC Rao, MD, Phd, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States